CLINICAL TRIAL: NCT00110669
Title: A Randomized Study of Daily vs. High-dose Weekly Prednisone Therapy in Duchenne Muscular Dystrophy
Brief Title: High-dose Prednisone in Duchenne Muscular Dystrophy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cooperative International Neuromuscular Research Group (Network)
Responsible Party: Study Chair, CINRG
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CNMC0601
Record Dates: First submitted 2005-05-12; First posted 2005-05-13 (Estimated); Last update posted 2011-10-27 (Estimated); Status verified 2011-10

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Muscular dystrophy, Duchenne and Beckers; Beckers Muscular dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Dystrophies | interventions — Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High Dose Prednisone (Active Comparator): Subjects who are randomized to the high-dose prednisone arm of the study will receive the following starting dose:
  •Prednisone at 10.0 mg/kg/wk (divided into two doses given on Saturday and Sunday)
  Interventions: Drug: Prednisone
- Daily Prednisone (Active Comparator): Subjects who are randomized to the daily prednisone arm of the study will receive the following starting dose:
  •Prednisone at 0.75 mg/kg/d
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Prednisone — Prednisone and dummy preparations for this study will be obtained from Frank's Pharmacy in Ocala, FL and will be supplied as a tablet containing 2.5mg, 5mg, 10mg, 20mg or 50mg Prednisone. Inactive "dummy" pills of similar look/taste will be supplied to maintain blinding.

SUMMARY:
This study will help to determine whether a high-dose weekly course of prednisone therapy is safer than and at least as effective as daily dose therapy for people with Duchenne muscular dystrophy (DMD). Boys who are enrolled in this study should not have taken carnitine, other amino acids, creatine, glutamine, Coenzyme Q10 or any herbal medicines within the last three months. There will be a two-visit screening to take place in one week to ensure a reproducible manual muscle test. The subject will then be randomized and put into either the daily or weekly regimen. The duration of the study is twelve 28-day treatment cycles (approximately 12 months) with follow-up visits at month one, three and then every three months.

DETAILED DESCRIPTION:
Duchenne muscular dystrophy (DMD) is the most common lethal inherited disorder worldwide. Despite the exponential increase in our understanding of the disorder since the discovery and characterization of the causative gene and its product dystrophin in 1987, current therapeutic management remains largely supportive. Awaiting a final genetic cure to be available in the future, further investments in developing better drug therapies for DMD remain important. The effect of a high dose prednisone regimen will be evaluated in comparison to a daily dose regimen in a multi-center, randomized, double-blind placebo-controlled 4-arm study. Ambulant children aged 4-10 years with an established DMD diagnosis will be studied. Patients will undergo 2 screening evaluations within 1 week. Patients will be randomized into treatment groups on the second screening visit, followed by a 12-month treatment period. During the treatment period, patients will be evaluated at monthly intervals. The primary endpoints are percentage change in average muscle strength score and QMT performance for specific muscle groups. Secondary endpoints include timed function tests, functional grades for arms and legs, and pulmonary function tests.

ELIGIBILITY:
Inclusion Criteria:

* 4 to 10 years of age
* Ambulant
* Confirmed DMD Diagnosis
* Steroid naive
* Evidence of muscle weakness by MRC score or clinical functional evaluation
* Ability to provide reproducible QMT bicep score

Exclusion Criteria:

* History of significant concomitant illness or significant impairment of renal or hepatic function, or other contraindication to steroid therapy
* Symptomatic DMD carrier
* Positive PPD
* Lack of prior exposure to chickenpox or immunization
* Use of carnitine, glutamine, Coenzyme Q10, other amino acids or any herbal medications within the last 3 months
* History of symptomatic cardiomyopathy
* Prior attainment of quota for the age group in which the patient belongs

Ages: 4 Years to 10 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2004-01; Primary Completion 2007-12 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Quantitative muscle strength will be measured using the CINRG Quantitative Measurement System (CQMS) | February 2008
Primary strength endpoints will be quantitative myometry (QMT) scores of the upper and lower extremities, consisting of paired flexor/extensor groups. | February 2008

SECONDARY OUTCOMES:
Secondary strength endpoints will include individual QMT scores of elbow and knee flexors and extensors and hand grip, manual muscle testing scores, which will be measured using the Medical Research Council's (MRC) muscle strength scoring method. | February 2008
Side-effect profiles will assessed by monitoring side-effects, including differences in growth (height and weight), calculated weight/height ratio, bone density, cataract formation, blood glucose, blood pressure and behavioral changes. | February 2008

CONTACTS AND LOCATIONS:
Overall Officials: Diana Escolar, MD, Study Chair — Children's National Research Institute
Locations (1):
- Children's National Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- See also: CINRG public website — http://www.cinrgresearch.org